CLINICAL TRIAL: NCT01229371
Title: Randomized, Parallel-group, Double-blind Multi-center Phase III Study to Assess the Immunogenicity and Safety of the 2010/2011-season Influenza Vaccine Formulated With Haemagglutinin (HA) Antigen From Two Suppliers, in Elderly and Young Adults
Brief Title: Immunogenicity and Safety Study to Assess Influenza Vaccine Formulated With Haemagglutinin (HA) Antigen From Two Suppliers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ADD-V-A001
Record Dates: First submitted 2010-10-22; First posted 2010-10-27 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Influenza; Virus; Vaccination; Immunisation
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects ≥18 to ≤60 Years - CSL HA Antigen (Active Comparator): Inflexal V influenza vaccine (CSL HA Antigen) 2010 Group A will be vaccinated with Inflexal V influenza vaccine (surface antigen, inactivated, virosome, using CSL HA Antigen) 2010/2011 containing per 0.5 mL i.m. dose: 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus; 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus; 15 μg HA antigen of B/Brisbane/60/2008-like virus
  Interventions: Biological: Inflexal V influenza vaccine (CSL HA Antigen) 2010
- Subjects >60 Years - CSL HA Antigen (Active Comparator): Inflexal V influenza vaccine (CSL HA Antigen) 2010 Group B will be vaccinated with Inflexal V influenza vaccine (surface antigen, inactivated, virosome, using CSL HA Antigen) 2010/2011 containing per 0.5 mL i.m. dose: 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus; 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus; 15 μg HA antigen of B/Brisbane/60/2008-like virus
  Interventions: Biological: Inflexal V influenza vaccine (CSL HA Antigen) 2010
- Subjects ≥18 to ≤60 Years - AdImmune HA Antigen (Experimental): Inflexal V influenza vaccine (AdImmune HA Antigen) 2010/2011 Group C will be vaccinated with Inflexal V influenza vaccine (surface antigen, inactivated, virosome, using AdImmune HA antigen) 2010/2011 containing per 0.5 mL i.m.dose: 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus; 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus; 15 μg HA antigen of B/Brisbane/60/2008-like virus
  Interventions: Biological: Inflexal V influenza vaccine (AdImmune HA antigen) 2010/2011
- Subjects >60 Years - AdImmune HA Antigen (Experimental): Inflexal V influenza vaccine (AdImmune HA Antigen) 2010/2011 Group D will be vaccinated with Inflexal V influenza vaccine (surface antigen, inactivated, virosome, using AdImmune HA antigen) 2010/2011 containing per 0.5 mL i.m.dose: 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus; 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus; 15 μg HA antigen of B/Brisbane/60/2008-like virus
  Interventions: Biological: Inflexal V influenza vaccine (AdImmune HA antigen) 2010/2011

INTERVENTIONS:
Biological: Inflexal V influenza vaccine (CSL HA Antigen) 2010 — Inflexal V influenza vaccine (surface antigen, inactivated, virosome, using CSL HA Antigen) 2010/2011, with intramuscular administration, containing per 0.5 mL dose: 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus; 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus; 15 μg HA antigen of B/Brisbane/60/2008-like virus
  Arms: Subjects >60 Years - CSL HA Antigen; Subjects ≥18 to ≤60 Years - CSL HA Antigen
Biological: Inflexal V influenza vaccine (AdImmune HA antigen) 2010/2011 — Inflexal V influenza vaccine (surface antigen, inactivated, virosome, using AdImmune HA antigen) 2010/2011 with intramuscular administration, containing per 0.5 mL dose: 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus; 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus; 15 μg HA antigen of B/Brisbane/60/2008-like virus
  Arms: Subjects >60 Years - AdImmune HA Antigen; Subjects ≥18 to ≤60 Years - AdImmune HA Antigen

SUMMARY:
The purpose of this study is to assess the humoral immune response and safety of the parenteral formulation of the 2010/2011-season virosomal subunit influenza vaccine Inflexal V using two different HA antigen suppliers (AdImmune and CSL), in groups of young and elderly adults, using the EMA (European Medicines Agency) regulation as a guideline.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the humoral immunogenicity and safety of the parenteral formulation of the 2010/2011-season influenza vaccine, Inflexal V, using HA antigen obtained from 2 different production facilities, and to compare the immunogenicity of both formulations to pre-defined EMA criteria for the annual relicensing of seasonal influenza vaccines. The evaluation will be done in young adults and elderly.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adults
* Aged ≥18 years on Day 1
* Written informed consent

Exclusion Criteria:

* Acute exacerbation of bronchopulmonary infection (cough, sputum, lung findings) or other acute disease
* Acute febrile illness (≥38.0 °C)
* Prior vaccination with an influenza vaccine (including the H1N1 pandemic swine flu vaccine) in the past 330 days
* Known hypersensitivity to any vaccine component
* Previous history of a serious adverse reaction to influenza vaccine
* History of egg protein allergy or severe atopy
* Known blood coagulation disorder
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of the study vaccine, incl. oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent (inhaled or topical steroids are allowed)
* Known immunodeficiency (incl. leukemia, cancer, HIV seropositivity)
* Investigational medicinal product received in the past 3 months (90 days)
* Treatment with immunoglobulins or blood transfusion(s) received in the past 3 months (90 days)
* Pregnancy or lactation
* Participation in another clinical trial
* Employee at the investigational site, or spouse and children of the investigator, or relative living in the same household as the investigator and/or are dependent on the investigator
* Suspected non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Seiberling, MD, Principal Investigator — Covance Clinical Research Unit AG
Locations (2):
- Switzerland (2):
  - Covance Clinical Research Unit AG, Allschwil
  - Cross Research S.A. Phase I Unit, Arzo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 19 October 2010 to 09 November 2010; outpatient study
Period: Overall Study
Arm/Group | Subjects ≥18 to ≤60 Years - AdImmune HA Antigen | Subjects ≥18 to ≤60 Years - CSL HA Antigen | Subjects >60 Years - AdImmune HA Antigen | Subjects >60 Years - CSL HA Antigen
Started | 109 | 111 | 110 | 110
Completed | 109 | 110 | 110 | 110
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects ≥18 to ≤60 Years - AdImmune HA Antigen | Subjects ≥18 to ≤60 Years - CSL HA Antigen | Subjects >60 Years - AdImmune HA Antigen | Subjects >60 Years - CSL HA Antigen | Total
Number analyzed (Participants) | 109 | 111 | 110 | 110 | 440
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 109 | 111 | 47 | 53 | 320
  >=65 years | 0 | 0 | 63 | 57 | 120
Age Continuous [Mean (Standard Deviation); unit: years] | 39.5 (11.18) | 39.9 (12.10) | 66.5 (5.50) | 66.4 (5.06) | 53.1 (16.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 50 | 49 | 53 | 206
  Male | 55 | 61 | 61 | 57 | 234
Region of Enrollment [Number; unit: participants]
  Switzerland | 109 | 111 | 110 | 110 | 440

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity - Geometric Mean Titer Fold Increase From Baseline
Description: The primary endpoints were the immunogenicity parameters for HA assessed via hemagglutinin inhibition method (HI). These parameters were analyzed according to the EMA "Note for guidance on harmonisation of requirements for influenza vaccines," 1997 and they were the following: 1. Seroprotection rate, defined as proportion of subjects with HI antibody titer ≥1:40, 2. Seroconversion rate, defined as proportion of subjects with ≥4-fold increase in HI antibody titer and with a titer of ≥1:40, 3. GMT of HI antibodies and fold-increase in GMT
Time Frame: 3 weeks after vaccination (Day 22 ± 2 days)
Population: Intent-to-treat population, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: GMT fold increase
Arm/Group | Subjects ≥18 to ≤60 Years - AdImmune HA Antigen | Subjects ≥18 to ≤60 Years - CSL HA Antigen | Subjects >60 Years - AdImmune HA Antigen | Subjects >60 Years - CSL HA Antigen
Number analyzed (Participants) | 109 | 110 | 110 | 110
GMT fold increase
  GMT fold increase from baseline: A/H1N1 | 3.5 [2.8 to 4.3] | 4.0 [3.3 to 5.0] | 4.5 [3.6 to 5.7] | 3.4 [2.8 to 4.2]
  GMT fold increase from baseline: A/H3N2 | 2.5 [2.1 to 3.0] | 2.5 [2.1 to 2.9] | 2.2 [1.8 to 2.6] | 1.9 [1.5 to 2.3]
  GMT fold increase from baseline: B-strain | 3.2 [2.6 to 3.8] | 3.1 [2.6 to 3.7] | 1.9 [1.7 to 2.2] | 2.1 [1.8 to 2.4]

2. Secondary Outcome: Number of Participants With Local and Systemic Adverse Events
Description: Solicited local and systemic AEs, Unsolicited AEs, Tolerability and acceptability
  Unsolicited AEs were collected from baseline (Day 1) to 3 weeks after vaccination (Day 22 ± 2 days).
  Solicited local and systemic AEs were collected by subjects diary from Day 1 (day of vaccination) to Day 4
Time Frame: Baseline (Day 1) and 3 weeks after vaccination (Day 22 ± 2 days)
Population: Safety population, all vaccinated subjects
Measure: Number; unit: participants
Arm/Group | Subjects ≥18 to ≤60 Years - AdImmune HA Antigen | Subjects ≥18 to ≤60 Years - CSL HA Antigen | Subjects >60 Years - AdImmune HA Antigen | Subjects >60 Years - CSL HA Antigen
Number analyzed (Participants) | 109 | 111 | 110 | 110
participants
  AEs (unsolicited and solicited) | 57 | 58 | 25 | 30
  Unsolicited AEs | 14 | 21 | 8 | 11
  Solicited local AEs | 45 | 41 | 18 | 21
  Solicited systemic AEs | 14 | 9 | 6 | 4

3. Primary Outcome: Immunogenicity - Seroprotection Rate
Description: as for outcome 1
Time Frame: 3 weeks after vaccination (Day 22 ± 2 days)
Population: Intent-to-treat population, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage subjects
Arm/Group | Subjects ≥18 to ≤60 Years - AdImmune HA Antigen | Subjects ≥18 to ≤60 Years - CSL HA Antigen | Subjects >60 Years - AdImmune HA Antigen | Subjects >60 Years - CSL HA Antigen
Number analyzed (Participants) | 109 | 110 | 110 | 110
percentage subjects
  Percentage of subjects seroprotected: A/H1N1 | 99.1 [95.0 to 100] | 98.2 [93.6 to 99.8] | 92.7 [82.8 to 96.8] | 90.0 [82.8 to 94.9]
  Percentage of subjects seroprotected: A/H3N2 | 99.1 [95.0 to 100] | 99.1 [95.0 to 100] | 100 [96.7 to 100] | 99.1 [95.0 to 100]
  Percentage of subjects seroprotected: B-strain | 96.3 [90.9 to 99.0] | 97.3 [92.2 to 99.4] | 85.5 [77.5 to 91.5] | 86.4 [78.5 to 92.2]

4. Primary Outcome: Immunogenicity - Seroconversion Rate
Description: as for outcome 1
Time Frame: 3 weeks after vaccination (Day 22 ± 2 days)
Population: Intent-to-treat population, vaccinated subjects with available pre- and post-vaccination titers
Measure: Number (95% Confidence Interval); unit: percentage subjects
Arm/Group | Subjects ≥18 to ≤60 Years - AdImmune HA Antigen | Subjects ≥18 to ≤60 Years - CSL HA Antigen | Subjects >60 Years - AdImmune HA Antigen | Subjects >60 Years - CSL HA Antigen
Number analyzed (Participants) | 109 | 110 | 110 | 110
percentage subjects
  Percentage of subjects seroprotected: A/H1N1 | 45.0 [35.4 to 54.8] | 52.7 [43.0 to 62.3] | 54.5 [44.8 to 64.1] | 43.6 [34.2 to 53.4]
  Percentage of subjects seroprotected: A/H3N2 | 27.5 [19.4 to 36.9] | 29.1 [20.8 to 38.5] | 25.5 [17.6 to 34.6] | 17.3 [10.7 to 25.7]
  Percentage of subjects seroprotected: B-strain | 40.4 [31.1 to 50.2] | 44.5 [35.1 to 54.3] | 20.9 [13.7 to 29.7] | 20.0 [13.0 to 28.7]

ADVERSE EVENTS:
Arm/Group | Subjects ≥18 to ≤60 Years - AdImmune HA Antigen | Subjects ≥18 to ≤60 Years - CSL HA Antigen | Subjects >60 Years - AdImmune HA Antigen | Subjects >60 Years - CSL HA Antigen
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/111 | 0/110 | 0/110
Other Adverse Events (participants affected / at risk) | 57/109 | 58/111 | 25/110 | 30/110
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects ≥18 to ≤60 Years - AdImmune HA Antigen (N=109) | Subjects ≥18 to ≤60 Years - CSL HA Antigen (N=111) | Subjects >60 Years - AdImmune HA Antigen (N=110) | Subjects >60 Years - CSL HA Antigen (N=110)
Chills (General disorders) | 7 (7) | 3 (3) | 4 (4) | 1 (1)
Fatigue (General disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Haemorrhage (at the injection site) (General disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Erythema (at the injection site) (General disorders) | 7 (7) | 6 (6) | 9 (9) | 5 (5)
Induration (at the injection site) (General disorders) | 11 (11) | 8 (8) | 9 (9) | 5 (5)
Pain (at the injection site) (General disorders) | 38 (38) | 39 (39) | 14 (14) | 14 (14)
Malaise (General disorders) | 12 (13) | 4 (4) | 6 (6) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period between 30 to 90 days (depending on the complexitiy of the work) from the time submitted to the sponsor for review.